CLINICAL TRIAL: NCT06367296
Title: Effects of a Resistance Exercise Training Program on Skeletal Muscle Quality, Immune Response and Physical Performance in Normal Weight Versus Obesity Older Women
Brief Title: Resistance Exercise Training in the Older Population With Obesity
Acronym: RETOPO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de La Frontera (Other)
Responsible Party: Principal Investigator, Nicolas Vidal-Seguel,, Principal Investigator, Universidad de La Frontera
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: RETOPO2024
Record Dates: First submitted 2024-04-02; First posted 2024-04-16 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Aging; Obesity
Keywords: Strength training; Malnutrition due to excess; Biochemical markers; Clinical anatomy
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal Weight (Experimental): All volunteers Normal Weight: BMI=18.5 kg/m2 to 24.9 kg/m2 and % fat <25.9%, n=16
  Interventions: Other: Prolonged resistance exercise training
- Obese (Experimental): All volunteers Obesity: BMI= 30.0 kg/m2 to 39.9 kg/m2 m2 and % fat > 32%, n=16.
  Interventions: Other: Prolonged resistance exercise training

INTERVENTIONS:
Other: Prolonged resistance exercise training — Training with resistance exercises for upper and lower limbs will be carried out 3 times a week (Monday, Wednesday and Friday) for 12 weeks for all participants. The training will follow the guidelines of the American College of Sports Medicine ("American College of Sports Medicine Position Stand. Progression Models in Resistance Training for Healthy Adults," 2009) and will consist of a 5-minute cardiovascular warm-up on a cycle ergometer, followed by weight training. Resistance training will be carried out with exercise machines: 5 sets of leg press, leg extension and leg flexion for lower limbs and 3 sets of chest press and triceps extension for upper limbs. Subsequently, the participants will perform global flexibility exercises for 5 minutes to return to calm.

SUMMARY:
Background:

Aging leads to an alteration in the immune response, characterized by a chronic inflammatory state, and a progressive decrease in muscle quantity and quality, a situation that increases in women and in the presence of obesity. With respect to muscle quality, intramuscular infiltration of adipose tissue has been considered a relevant parameter, involved in the relationship between aging-obesity-inflammation. As a therapeutic strategy, physical training with resistance exercises (or also known as strength training) has been shown to be effective in increasing skeletal muscle mass in this age group. However, its role on muscle quality in normal-weight versus obese older women has not been fully addressed.

Hypothesis:

A 12-week resistance exercise training program is effective in improving muscle quality, immune response and physical performance in normal weight and obese older women. In addition to the above, the investigators hypothesize that women with obesity will present greater baseline alterations, so the percentage of change will be higher compared to older women with normal weight after the training program.

Goals:

The primary aim of this study is to evaluate the effects of a 12-week resistance exercise training on muscle quality (infiltration of intramuscular adipose tissue), immune response and physical performance in older women between 60 and 79 years of age with obesity compared to older women with normal weight of the same age range.

Methodology:

The present clinical trial will consider 2 groups of older women between 60 and 79 years old: normal weight (BMI=18.5 to 24.9 kg/m 2 and % fat <25.9) and obese (BMI =30 to 39.9 Kg/m 2 and fat % >32). Participants will perform 12 weeks of training with resistance exercises 3 times a week. Before and after training, intramuscular infiltration of adipose tissue (echogenicity) will be measured by ultrasound, followed by aspects of muscle architecture (muscle thickness, penile angle and fascicle length) and functional parameters of muscle quality (maximum strength determined by 1 repetition maximum-1RM, maximum voluntary isometric strength of knee extensors through a lower limb force and power transducer). Finally, fasting blood samples will be obtained (immune response) and physical performance, body composition, physical activity level, and quality of life will be evaluated.

DETAILED DESCRIPTION:
Background:

Aging leads to an alteration in the immune response, characterized by a chronic inflammatory state, and a progressive decrease in muscle quantity and quality, a situation that increases in women and in the presence of obesity. With respect to muscle quality, intramuscular infiltration of adipose tissue has been considered a relevant parameter, involved in the relationship between aging-obesity-inflammation. As a therapeutic strategy, physical training with resistance exercises (or also known as strength training) has been shown to be effective in increasing skeletal muscle mass in this age group. However, its role on muscle quality in normal-weight versus obese older women has not been fully addressed.

Hypothesis:

A 12-week resistance exercise training program is effective in improving muscle quality, immune response and physical performance in normal weight and obese older women. In addition to the above, the investigators hypothesize that women with obesity will present greater baseline alterations, so the percentage of change will be higher compared to older women with normal weight after the training program.

Goals:

The primary aim of this study is evaluate the effects of a 12-week resistance exercise training on muscle quality (infiltration of intramuscular adipose tissue), immune response and physical performance in older women between 60 and 79 years of age with obesity compared to older women with normal weight of the same age range.

Specific goals:

To evaluate the effects of a 12-week resistance exercise training program in elderly women between 60 and 79 years of age with obesity, in comparison to older people with normal weight of the same age range on parameters of:

* Muscle architecture (muscle thickness, pennation angle and fascicle length) and muscle quality functionalities (power and strength).
* Immune response through inflammatory cytokines: Tumor necrosis factor a (TNFa) interleukin-1 (IL-1), IL-6, IL-8 and induction of neutrophil extracellular traps (NETosis).
* Physical performance (SPPB), Body composition (BIA) and quality of life (SF-36).

Methodology:

The present clinical trial will consider 2 study groups of older women between 60 and 79 years old: normal weight (BMI=18.5 to 24.9 kg/m 2 and % fat <25.9) and obese (BMI =30 to 39.9 Kg/m 2 and fat % >32). Participants will perform 12 weeks of training with resistance exercises 3 times a week. Before and after training, intramuscular infiltration of adipose tissue (echogenicity) will be measured by ultrasound, followed by aspects of muscle architecture (muscle thickness, penile angle and fascicle length) and functional parameters of muscle quality (maximum strength determined by 1 repetition maximum-1RM, maximum voluntary isometric strength of knee extensors through a lower limb force and power transducer). Finally, fasting blood samples will be obtained (immune response) and physical performance, body composition, physical activity level, and quality of life will be evaluated.

Study parameters/endpoints

* The main study endpoint is the decrease in echointensity as a marker of muscle quality, evaluated through ultrasonography in the quadriceps muscles of the lower limbs of participants subjected to 12 weeks of resistance training.
* Secondary endpoints include: Muscle architecture parameter (morphological aspects of muscle quality); muscle thickness, pennation angle and fascicle length; Functional parameters of muscle quality, maximum voluntary isometric strength of knee extensors and lower limb power; Immune response in blood (TNFa, IL-1, IL-6, IL-8 and NETosis); Physical performance (SPPB), evaluation of maximum strength (1RM) and handgrip strength; Body composition (fat mass and total muscle mass and for each lower limb) and anthropometry (waist - hip, thigh and calf circumference, leg length and knee height); And Level of physical activity (IPAQ) and Quality of Life (SF-36).
* Other study parameters include: Age, body weight, body height, body mass index (BMI), lipid profile, glucose, insulin, HOMA index, blood pressure, heart rate and perception of effort using the Borg scale.

Expected results:

The effect of resistance exercise training on muscle quality in normal-weight versus obese older women is still unclear. The present research project aims to demonstrate the effectiveness of this training modality in improving muscle quality parameters, as well as measures of immune response and physical performance in older women. However, the investigators believe that the impact will be greater in women with obesity, as they present greater baseline alterations compared to older normal weight women. The possible findings will define the scientific-practical foundations for the prescription of physical training in older women with obesity.

ELIGIBILITY:
Inclusion Criteria:

* Older women between 60 and 79 years old who live in the community, that is, they do not live in nursing homes or similar.
* Older people with normal weight (BMI=18.5 to 24.9 kg/m2 and % fat <25.9) and those with obesity (BMI= 30 to 39.9 Kg/m2 and % fat > 32).
* Cognitive ability to follow verbal orders.

Exclusion Criteria:

* Neuromuscular or mobility disorders that do not allow resistance training to be carried out safely (debilitating arthritis, spasticity/rigidity, neurological disorders and paralysis).
* Use of nutritional supplementation that can regulate skeletal muscle (leucine, glutamine, casein, whey-protein, fatty acids and creatine).
* Untreated and/or uncontrolled chronic diseases.
* Have carried out a training program with resistance exercises in the last 6 months.

Ages: 60 Years to 79 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-01-28 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in intermuscular adipose tissue (measured via ultrasonography) after prolonged resistance-type exercise training | Before, and after 12 weeks of training
  Intramuscular adipose tissue infiltration evaluated by echointensity (Pixel Intensity 0 to 255) in the rectus femoris and vastus intermedius muscles of both lower limbs

SECONDARY OUTCOMES:
Change in muscle thickness (measured via ultrasonography) after prolonged resistance-type exercise training | Before, and after 12 weeks of training
  Muscle thickness (centimeters) evaluated in the rectus femoris and vastus intermedius muscles of both lower limbs. The muscle thickness evaluated as the distance between the deep and superficial fascia.
Change in pennation angle (measured via ultrasonography) after prolonged resistance-type exercise training | Before, and after 12 weeks of training
  Pennation angle (degree) evaluated in the rectus femoris and vastus intermedius muscles of both lower limbs. The pennation angle evaluated as the angle between the fascicle and the deep fascia. The average of three measurements will be calculated
Change in fascicle length (measured via ultrasonography) after prolonged resistance-type exercise training | Before, and after 12 weeks of training
  Fascicle length (centimeters) evaluated in the rectus femoris and vastus intermedius muscles of both lower limbs. Fascicle length = sin(y +90º) × MT/ sin(180º-(y +180º- PA)), where "y" is the angle between the superficial and deep facia, while PA is the pennation angle, while MT is the Muscle thickness.
Change in physical performance (measured via Short physical performance battery (SPPB)) after prolonged resistance-type exercise training | Before, and after 12 weeks of training
  Measurement of physical performance via SPPB
Change in arms and legs strength (measured via 1-Repetition Maximum (1RM) testing) after prolonged resistance-type exercise training | Before, and after 12 weeks of training
  Maximal strength assessment via 1RM testing of leg press, leg extension, leg flexion, chest press and triceps extension
Change in hand grip strength (measured via JAMAR(R) handheld dynamometer) after prolonged resistance-type exercise training | Before, and after 12 weeks of training
  Maximal strength assessment via 1RM testing of JAMAR(R) handheld dynamometer.
Change in maximum voluntary isometric strength (measured via Force transducer) after prolonged resistance-type exercise training. | Before, and after 12 weeks of training
  The maximum voluntary isometric knee extension force (Newton) evaluated in both lower limbs (always maintaining randomness in the limbs).
Change in muscle power of the lower limbs (measured via Five Times Sit to Stand test) after prolonged resistance-type exercise training. | Before, and after 12 weeks of training
  The muscle power of the lower limbs (Watt) evaluated by equation STS Men Power.
Change in Immune response in blood (measured via flow cytometry) after prolonged resistance-type exercise training. | Before, and after 12 weeks of training
  The immune response evaluated by TNFa,IL-1, IL-6, IL-8 (pg/ml)
Change in NETosis in blood (measured via IncuCyte) after prolonged resistance-type exercise training. | Before, and after 12 weeks of training
  The NETosis (%) evaluated with live cell imaging in donated neutrophils cultured with serum from the participants for 30 h.
Change in Whole body lean mass (measured via Bioimpedance) after prolonged resistance-type exercise training. | Before, and after 12 weeks of training
  The Whole Body lean mass (Kg) through TANITA MC 980U PLUS
Change in Whole body fat mass (measured via Bioimpedance) after prolonged resistance-type exercise training. | Before, and after 12 weeks of training
  The Whole Body fat mass (Kg) through TANITA MC 980U PLUS
Change in Physical activity level (measured via IPAQ short version) after prolonged resistance-type exercise training. | Before, and after 12 weeks of training
  The physical activity level evaluated by International Physical Activity Questionnaire, short version. Classifying the level of physical activity as low, moderate or high.
Change in Quality of Life level (measured via SF-36) after prolonged resistance-type exercise training. | Before, and after 12 weeks of training
  The Quality of Life level evaluated by SF-36 questionnaire. The score ranges from 0 to 100%, where a higher score High implies a better quality of life related to health.

CONTACTS AND LOCATIONS:
Overall Officials: GABRIEL MARZUCA, Msc, PhD, Study Director — Universidad de La Frontera. Temuco, Chile
Locations (2):
- Chile (2):
  - Universidad de La Frontera, Temuco, IX Región de La Araucanía
  - Gabriel Marzuca, Temuco, Región de la Araucanía

IPD SHARING:
Plan to Share IPD: No